CLINICAL TRIAL: NCT01189734
Title: Comparison Between Laparoscopic Common Bile Duct Exploration and Intraoperative ERCP for Management of Common Bile Duct Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LCBDEIOES
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-02

CONDITIONS: Common Bile Duct Gallstones
Keywords: common bile duct stones; laparoscopic common bile duct exploration; intraoperative ercp; Preoperatively diagnosed common bile duct stones
MeSH Terms: conditions — Gallstones | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- laparoscopic common bile duct exploration (Placebo Comparator)
  Interventions: Procedure: laparoscopic common bile duct exploration
- laparoscopic cholecystectomy with intraoperative ES (Active Comparator)
  Interventions: Procedure: laparoscopic cholecystectomy and intraoperative endoscopic sphincterotomy

INTERVENTIONS:
Procedure: laparoscopic common bile duct exploration
  Arms: laparoscopic common bile duct exploration
Procedure: laparoscopic cholecystectomy and intraoperative endoscopic sphincterotomy
  Arms: laparoscopic cholecystectomy with intraoperative ES

SUMMARY:
Many options are available for management of common bile duct stones. the most recent development in this field is single-session approach by one of two methods; laparoscopic common bile duct exploration and intraoperative endoscopic sphincterotomy. In this study, the investigators prospectively compare these two methods for management of patients with preoperatively diagnosed common bile duct stones to settle the best option.

ELIGIBILITY:
Inclusion Criteria:

* preoperatively diagnosed common bile duct stones

Exclusion Criteria:

* liver cirrhosis pregnancy ASA III, IV Previous abdominal surgery postcholecystectomy

Ages: 12 Years to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 248 (Actual)

PRIMARY OUTCOMES:
success/failure of common bile duct removal

SECONDARY OUTCOMES:
Surgical time

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Surgical Center, Al Mansurah, Dakahlia Governorate, Egypt